CLINICAL TRIAL: NCT03383640
Title: Will Early Active Finger Exercises in Replanted Fingers Improve Mobility? A Prospective Randomized Trial
Brief Title: Early Active Finger Exercises in Replanted Fingers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johanne Korslund, Doctor, orthopaedic surgeon, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1282 D
Record Dates: First submitted 2017-12-15; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control Group: Standardized post operative rehabilitation, where active exercises of the replanted digits is postponed until radiologic healing of the amputated bone.
- Intervention (Other): Intervention Group: Early active exercises of the replanted digits started between day 5 and 7 after surgery, as instructed by hand therapist
  Interventions: Other: Active exercises

INTERVENTIONS:
Other: Active exercises — Active flexion movements every waking hour of the replanted digits
  Arms: Intervention

SUMMARY:
A controlled randomized trial, including patients undergoing finger replantation surgery. The Control Group will receive a standardized post operative rehabilitation regime, whilst the Intervention Group will receive a rehabilitation regime that includes early active exercises of the replanted digits.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Total or subtotal amputation injury of 1-4 of the four ulnar digits
* Injury distal to the MCP joint
* Must have injured flexor tendon which requires suture
* Must have a fracture
* Surgery done with a stable osteosynthesis with acceptable post-operative x-ray imaging
* The finger must have had a stable circulation for at least 5 days post-surgery

Exclusion Criteria:

* Arthrodesis/temporary fixation of the MCP joint
* Bilateral amputation injury
* Severely damage of other parts if the hand compromising the patient's ability to perform active exercises of the fingers
* Patients who cannot follow the planned controls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-05 (Estimated)

PRIMARY OUTCOMES:
TAM | 12 months
  Total active movement of the interphalangeal joints

SECONDARY OUTCOMES:
Quick-DASH | 12 months
  Upper extremity function score (patient related outcome measure)
VAS Pain | 12 months
  Visual Analogue Score Pain
VAS Function | 12 months
  Visual Analogue Score Function
Grip strength | 12 months
  Jamar dynanometer
Key pinch | 12 months
  Jamar dynamometer